CLINICAL TRIAL: NCT02292524
Title: Prostate Biomarkers in Men Consuming Tomato Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Schwartz, Steven, PhD (Unknown)
Responsible Party: Principal Investigator, Steven Clinton, Steven Clinton, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-0137
Record Dates: First submitted 2014-10-31; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I: Control (No Intervention): Men in this group consumed a tomato free diet for the duration of the study (less than or equal to 5 mg lycopene/day) and, thus, did not consume a tomato intervention product.
- Arm II: Juice (Experimental): Commercially-available tomato food product: men in this group consumed V8® juice (11-16.5 fl. oz./day).
  Interventions: Other: Commercially-available tomato food product
- Arm III: Soup (Experimental): Commercially-available tomato food product: men in this group consumed Campbell's® Tomato Soup (2-2 ¾ cups/day).
  Interventions: Other: Commercially-available tomato food product
- Arm IV: Sauce (Experimental): Commercially-available tomato food product: men in this group consumed Prego® spaghetti sauce (5-7 oz./day).
  Interventions: Other: Commercially-available tomato food product

INTERVENTIONS:
Other: Commercially-available tomato food product — Each of the three tomato food products (juice, soup, sauce) provided 25-35 mg lycopene/day.
  Arms: Arm II: Juice; Arm III: Soup; Arm IV: Sauce

SUMMARY:
Prostate Biomarkers in Men Consuming Tomato Products

DETAILED DESCRIPTION:
Participants completed a minimum week-long washout period without consumption of tomato products prior to randomization to one of four dietary interventions. Men were randomized to one of the following dietary interventions: a controlled low lycopene diet (≤ 5 mg/d from foods), daily Prego® spaghetti sauce, daily V8® vegetable juice, or daily Campbell's® Tomato Soup. Each of the tomato products provided between 25 and 35 mg lycopene per day. In order to provide this dietary intervention in typical serving sizes in the context of a usual diet but devoid of other tomato sources, participants kept daily logs documenting compliance with the intervention product and a tomato-restricted diet from enrollment to the day of surgery (~3 weeks). Study participants were asked to complete an abbreviated dietary history questionnaire (to establish typical consumption patterns of various tomato products) and two separate 3-day diet food records, once during the washout and once during the intervention period. Blood and 24-hour urine samples were obtained at two time points, after the one-week washout phase and at the end of the dietary intervention period. Fresh prostate samples were obtained at time of surgery.

ELIGIBILITY:
Inclusion Criteria: To be included in this study, men must:

* Have biopsy-proven, clinically localized adenocarcinoma of the prostate based on standard presurgical staging studies
* Have chosen to undergo a radical prostatectomy for treatment of their disease after the medical team has presented all possible treatment options
* Have kidney and liver enzymes, CBC, and PT/PTT/INR within normal limits
* Agree to sign consent form prior to enrollment in the study

Exclusion Criteria: Men may not participate in this if they:

* Are currently taking lycopene or "alternative" dietary supplements
* Have a history of digestive or malabsorptive disorders, metabolic enzyme deficiencies, or other disorders requiring special dietary modifications (controlled type II diabetes mellitus was allowed)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-05; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Measure carotenoids, including lycopene and its isomers, in blood (umol/L) and prostate tissue (nmol/g) of men after three weeks of consuming V8 vegetable juice, condensed tomato soup or tomato sauce. | Day 0 and End of Study (an average of 23 days)

SECONDARY OUTCOMES:
Measure histobiomarkers in the prostate related to aggressive disease including Gleason Grade (number 1 - 10), tumor volume (weight) , and vascular endothelial growth factor expression (ng/mL) | Day 0 and End of Study (an average of 23 days)
  Measure histobiomarkers in the prostate related to aggressive disease including Gleason Grade, tumor volume, and vascular endothelial growth factor expression
Measure biomarkers related to prostate cancer in controls and men consuming tomato food products prior to surgery. These biomarkers include plasma insulin like growth factor (ng/mL) and plasma prostate specific antigen (ng/mL) | Day 0 and End of study (an average of 23 days)
  Measure biomarkers related to prostate cancer in controls and men consuming tomato food products prior to surgery. These biomarkers include plasma insulin like growth factor (ng/mL) and plasma prostate specific antigen (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center/ We, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu